CLINICAL TRIAL: NCT01962350
Title: Evaluation Clinical, Cognitive and Safety in the Treatment of Bipolar Depression With H1-Coil Deep Transcranial Magnetic Stimulation
Brief Title: Treatment of Bipolar Depression With H1-Coil Deep Brain rTMS: Clinical-Cognitive and Safety Evaluation
Acronym: rTMSH1Coil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, Andre Brunoni, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 150.067/12
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Bipolar Depression
Keywords: Deep Brain Transcranial Magnetic Stimulation;; H1-Coil deep brain rTMS;; H1-Coil;; Bipolar Depression;; Cognition.
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active H1-Coil deep brain rTMS (Experimental): Deep Brain Transcranial Magnetic Stimulation
  18Hz Active H1-Coil deep brain rTMS for 4-weeks over the cortex prefrontal. n=25
  Interventions: Device: Deep Brain Transcranial Magnetic Stimulation
- Sham H1-Coil deep brain rTMS (Experimental): Deep Brain Transcranial Magnetic Stimulation
  Sham H1-Coil deep brain rTMS for 4-weeks over the cortex prefrontal. n=25
  Interventions: Device: Deep Brain Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Deep Brain Transcranial Magnetic Stimulation — H1-Coil deep brain rTMS at cortex prefrontal.
  Other Names: H1-Coil deep brain rTMS;; H1-Coil.

SUMMARY:
The treatment of bipolar disorders is always a challenge in daily practice. Mood stabilizers are partially effective in the treatment of depressive phase of the illness, although there are some reports relating to the antidepressant properties of these drugs. Other conventional methods (pharmacological) and non- conventional treatment are not effective or involve risks and side effects. Several studies with Transcranial Magnetic Stimulation (TMS) showed that magnetic stimulation daily over the left prefrontal cortex may improve the mood of patients. TMS is a noninvasive method of stimulating the brain. The instrument used nowadays in local research and application Clinical is a metallic coil formed in figure 8 (coil format 8). This instrument was capable of stimulating only surface areas of the brain, primarily the cerebral cortex, at depths of up to 3 inches below the scalp. From this angle, there is clearly a need for a means of producing magnetic fields which can reach deeper brain areas, such as those involved in mood disorders. TMS has little, if any effect in these brain areas. To this end, new coils, calls "H", that promote the stimulation of deep brain areas were developed in collaboration with the National Institute of Health (NIH) in the USA. This new coil - H1 that will be evaluated in this study has been tested for safety in NIH in 2003 by Dr. Abraham Zangen. Yet there are very few prospective clinical, randomized and controlled trials, on the effects of early and late in clinical-cognitive condition and safety of TMS with H1 coils in treating episodes of bipolar depression. The application of EMT with H1 coils can reach deepest regions of the brain and improve the clinical and cognitive condition of subjects with episodes of bipolar depression, and may be confirmed as a safe and virtually free of side effects. By an absence of treatment actually effective for bipolar depression, this study will show whether there are clinical and cognitive benefits of deep TMS with H1 coil in patients with bipolar depression.

DETAILED DESCRIPTION:
The present research protocol will evaluate clinical-cognitive and safety effects of H1-Coil Deep Brain Transcranial Magnetic Stimulation over prefrontal cortex in subjects with bipolar depression, currently treated with mood stabilizer and/or antipsychotics for stabilization and sleep regulation. Patients will be clinically evaluated with the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) criteria for Bipolar Depressive Episode. Symptoms intensity will be rated according to The Hamilton Depression Scale (HAMD -17 items) - main outcome. Patients with scores higher than 18 will be included and the cognitives functions will be evaluated according with tasks of neuropsychologic battery chosen. Patients with active neurological or severe disorders (such as cancer, auto-imune and cardiologic disorders) will be excluded. The present study is a double-blinded, controlled, randomized trial with 50 patients in bipolar depression episode. The intervention protocol consist in 20 consecutive daily deep TMS sessions (skipping the weekend). After meeting eligibility criteria, patients will be randomized (computer generated list) to one of the two intervention groups: 25 patients in Active H1-Coil deep brain rTMS group and Sham H1-Coil deep brain rTMS group. H1-Coil deep brain rTMS sessions will follow the following steps: the first day of treatment, patients will be instructed to wear earplugs to minimize the risk of impaired hearing. Then, the threshold intensity of stimulation motor is determined by applying pulses only to the motor cortex. The stimulation threshold is determined pro gradually increase the stimulation intensity every 5 seconds. The stimulation threshold is defined as stimulation of lesser intensity that can evoked motor potential with at least 50μV amplitude of at least 5 tentativas.A coil is positioned to 5 centimeters below the hot spot (in the prefrontal area) intensity - 120% of the threshold engine. Each session will receive 55 groups of stimuli, duration - 2/2 , frequency - 18 Hz , area - left prefrontal , intervals - 20 seconds . Soon, 1,980 pulses of magnetic stimulation will be administered every day (per session), totaling 39,600 pulses throughout treatment. Patients will be clinically assessed at baseline, weekly during the four weeks of treatment and for four weeks after completion of treatment ending in 8 weeks. Main outcome will be based on HAMD-17 items at a endpoint of 4-weeks and follow up 4-weeks, with secondary outcomes assessing Young Mania Rating Scale (11 items) at 8 weeks. Other evaluation scales include, Hamilton Anxiety Scale, Global Assessment Scale and Clinical Global Impression at 8 weeks. The cognitive assessment will be performed with a neuropsychologic battery tests at baseline, endpoint of 4-weeks and endpoint of 8-weeks with a trained neuropsychologist. Also a Safety Deep rTMS Scale, adverse effects scales and clinical evaluation with a trained physician.

ELIGIBILITY:
Inclusion Criteria: Outpatients

* Diagnosed by two senior psychiatrists as suffering from bipolar depression (BP1, BP2) episode according to DSM IV using the Structured Clinical Interview for DSM-4 (SCID), with additional requirement of duration for the current episode ≥ 4 weeks and CGI ≥ 4.
* First Stimulation threshold: intensity ≤ 70% of the threshold engine.
* Rating on HAM-D (17 items) >18 at the screening visit.
* Age: 18-65 years.
* Gave informed consent for participation in the study.
* Negative answers on safety screening questionnaire for transcranial magnetic stimulation
* Taking mood stabilizing medication (e.g., lithium) on an acceptable range of dosage according to recent blood examination or antipsychotic medication as mood stabilizers prescribed by their treating physician
* According to the treating physician the patient is compliant in taking the mood-stabilizing medication.
* Medication resistance to at least two different antidepressant treatments, defined as resistance to a minimum of 2 antidepressant drug trials of adequate dose and duration in the current episode or previous episodes defined as a minimum level of 3 on the ATHF per antidepressant drug-trial.
* Patients who have not completed antidepressant trials of adequate dose and duration due to intolerance to therapy may be included if they have demonstrated intolerance to 3 or more anti-depressant medications in the current or a previous episodes.
* If currently taking antidepressant pharmacotherapy, must be clinically appropriate to discontinue treatment with those agents.
* Able to tolerate psychotropic medication washout and no psychotropics during the H-coil deep brain rTMS other than benzodiazepine at equivalent dose of up to 3 mg lorazepam every day.
* Right hand dominance.

Exclusion Criteria: Diagnosis as suffering from other diagnosis on axis 1 (like: schizophrenia, geriatric depression).

* Diagnosis as suffering from Severe Borderline Personality Disorder or hospitalized due to exacerbation related to of borderline personality disorder.
* Substantial suicidal risk as judged by the treating psychiatrist.
* Attempted suicide in the past year.
* Patients with a bipolar cycle of less than 30 days.
* History of epilepsy or seizure in first degree relatives.
* History of head injury.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of frequent or severe headaches.
* History of migraine.
* History of hearing loss.
* Known history of cochlear implants.
* History of substance abuse within the past 6 months (except nicotine and caffeine) or alcoholism.
* Pregnancy or not using a reliable method of birth control.
* Unstable Systemic and metabolic disorders.
* Unstable neurological or medical disease.
* Inadequate communication with the patient.
* Under custodial care.
* Participation in current clinical study or clinical study within 30 days prior to this study.
* Participants who suffer from an unstable physical disease such as high blood pressure or acute, unstable cardiac disease
* Use of fluoxetine within 6 weeks of the baseline visit
* Use of a Monoamine Oxidase Inhibitor (MAOI) within 2 weeks of the baseline visit
* Current use of antidepressant medications during the course of the trial.
* Current use of Leponex (Clozapine).
* Previous treatment with TMS
* Women who are breast-feeding
* Known or suspected pregnancy
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression, 17 items (HAMD17) | Weeks 0, 4 and 8
  Reduction of depressive symptoms as assessed by HAMD17

SECONDARY OUTCOMES:
Young Mania Rating Scale (11 items) | During the eight weeks
  safety: to control manic symptoms.

OTHER OUTCOMES:
Neuropsychologic Battery Tasks | week 0, 4 and 8
  A set of tests for cognitive functions such as attention, memory, mental flexibility, processing speed, reaction time, visuo-spacial perception, executive functions and language that, often show deficits in patients with bipolar depression.

CONTACTS AND LOCATIONS:
Overall Officials: Andre B Brunoni, Phd, Study Director — Department and Institute of Psychiatry, General Hospital, University of Sao Paulo Medical School
Locations (1):
- Department of Psychiatry - University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rosenberg O, Isserles M, Levkovitz Y, Kotler M, Zangen A, Dannon PN. Effectiveness of a second deep TMS in depression: a brief report. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Jun 1;35(4):1041-4. doi: 10.1016/j.pnpbp.2011.02.015. Epub 2011 Feb 24. PMID 21354242
- [Background] Rosenberg O, Roth Y, Kotler M, Zangen A, Dannon P. Deep transcranial magnetic stimulation for the treatment of auditory hallucinations: a preliminary open-label study. Ann Gen Psychiatry. 2011 Feb 9;10(1):3. doi: 10.1186/1744-859X-10-3. PMID 21303566
- [Background] Rosenberg O, Zangen A, Stryjer R, Kotler M, Dannon PN. Response to deep TMS in depressive patients with previous electroconvulsive treatment. Brain Stimul. 2010 Oct;3(4):211-7. doi: 10.1016/j.brs.2009.12.001. Epub 2009 Dec 30. PMID 20965450
- [Background] Rosenberg O, Shoenfeld N, Zangen A, Kotler M, Dannon PN. Deep TMS in a resistant major depressive disorder: a brief report. Depress Anxiety. 2010 May;27(5):465-9. doi: 10.1002/da.20689. PMID 20455247
- [Background] Levkovitz Y, Roth Y, Harel EV, Braw Y, Sheer A, Zangen A. A randomized controlled feasibility and safety study of deep transcranial magnetic stimulation. Clin Neurophysiol. 2007 Dec;118(12):2730-44. doi: 10.1016/j.clinph.2007.09.061. Epub 2007 Oct 30. PMID 17977787
- [Background] Roth Y, Amir A, Levkovitz Y, Zangen A. Three-dimensional distribution of the electric field induced in the brain by transcranial magnetic stimulation using figure-8 and deep H-coils. J Clin Neurophysiol. 2007 Feb;24(1):31-8. doi: 10.1097/WNP.0b013e31802fa393. PMID 17277575
- [Background] Poon SH, Sim K, Sum MY, Kuswanto CN, Baldessarini RJ. Evidence-based options for treatment-resistant adult bipolar disorder patients. Bipolar Disord. 2012 Sep;14(6):573-84. doi: 10.1111/j.1399-5618.2012.01042.x. PMID 22938165
- [Background] Bersani FS, Minichino A, Enticott PG, Mazzarini L, Khan N, Antonacci G, Raccah RN, Salviati M, Delle Chiaie R, Bersani G, Fitzgerald PB, Biondi M. Deep transcranial magnetic stimulation as a treatment for psychiatric disorders: a comprehensive review. Eur Psychiatry. 2013 Jan;28(1):30-9. doi: 10.1016/j.eurpsy.2012.02.006. Epub 2012 May 3. PMID 22559998
- [Background] Loo C, Katalinic N, Mitchell PB, Greenberg B. Physical treatments for bipolar disorder: a review of electroconvulsive therapy, stereotactic surgery and other brain stimulation techniques. J Affect Disord. 2011 Jul;132(1-2):1-13. doi: 10.1016/j.jad.2010.08.017. Epub 2010 Sep 21. PMID 20858566
- [Background] Richieri R, Adida M, Dumas R, Fakra E, Azorin JM, Pringuey D, Lancon C. [Affective disorders and repetitive transcranial magnetic stimulation: Therapeutic innovations]. Encephale. 2010 Dec;36 Suppl 6:S197-201. doi: 10.1016/S0013-7006(10)70057-9. French. PMID 21237356
- [Result] Bersani FS, Girardi N, Sanna L, Mazzarini L, Santucci C, Kotzalidis GD, Sani G, De Rossi P, Raccah RN, Caltagirone SS, Battipaglia M, Capezzuto S, Bersani G, Girardi P. Deep transcranial magnetic stimulation for treatment-resistant bipolar depression: a case report of acute and maintenance efficacy. Neurocase. 2013;19(5):451-7. doi: 10.1080/13554794.2012.690429. Epub 2012 Jul 24. PMID 22827578
- [Result] Harel EV, Zangen A, Roth Y, Reti I, Braw Y, Levkovitz Y. H-coil repetitive transcranial magnetic stimulation for the treatment of bipolar depression: an add-on, safety and feasibility study. World J Biol Psychiatry. 2011 Mar;12(2):119-26. doi: 10.3109/15622975.2010.510893. Epub 2010 Sep 21. PMID 20854181